CLINICAL TRIAL: NCT03648762
Title: Exercise Therapy to Reduce Heart Failure Symptoms; Sorting Mechanisms of Benefit
Acronym: EXT-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: O0834-R
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Results first posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure
Keywords: Heart failure; Exercise; Cardiopulmonary
MeSH Terms: conditions — Heart Failure; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants with heart failure will complete 1 of 3 exercise training interventions (aerobic vs. aerobic and strength vs. inspiratory) for 12 weeks and will be assessed pre and post to determine if any differences occur in their skeletal muscle and functional capacity as part of the exercise intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Aerobic Exercise Intervention (Other): 12 weeks of a minimum of 3 days a week for 60 minutes of aerobic exercise
  Interventions: Behavioral: Aerobic Exercise Intervention
- Combined Aerobic and Strength Exercise Intervention (Other): 12 weeks of a minimum of 3 days a week for 60 minutes of Combined Aerobic and Strength Exercise
  Interventions: Behavioral: Combined Aerobic and Strength Exercise Intervention
- Inspiratory Muscle Training Exercise Intervention (Other): 12 weeks of a minimum of 3 days a week for 60 minutes of Inspiratory Muscle Training Exercise
  Interventions: Behavioral: Inspiratory Muscle Training Exercise Intervention

INTERVENTIONS:
Behavioral: Aerobic Exercise Intervention — Aerobic Exercise Intervention - 12 weeks of a minimum of 3 days a week for 60 minutes of aerobic exercise
  Arms: Aerobic Exercise Intervention
Behavioral: Combined Aerobic and Strength Exercise Intervention — Combined Aerobic and Strength Exercise Intervention- 12 weeks of a minimum of 3 days a week for 60 minutes of Combined Aerobic and Strength Exercise
  Arms: Combined Aerobic and Strength Exercise Intervention
Behavioral: Inspiratory Muscle Training Exercise Intervention — Inspiratory Muscle Training Exercise Intervention- 12 weeks of a minimum of 3 days a week for 60 minutes of Inspiratory Muscle Training Exercise
  Arms: Inspiratory Muscle Training Exercise Intervention

SUMMARY:
The purpose of this research study is to better understand how exercise training in older adults (≥65 years) with heart failure (HF) affects skeletal muscle both intrinsically and in respect to its impact on functional capacity. While many conceptualize HF as a pathophysiology that exclusively affects the heart, skeletal muscle atrophy and weakening are also elemental to the disease. While reduced exercise capacity is typically associated with HF, this may be related more to disease effects in skeletal muscle than the heart. This is a clinical study that focuses on exercise training which compares functional endpoints before and after training. Patients are randomized to one of three exercise training interventions (aerobic vs. aerobic and strength vs. inspiratory muscle training) for 12 weeks and are assessed pre- and post-training to determine if any differences occur in their skeletal muscle and functional capacity. Skeletal muscle biopsies before and after the exercise training intervention in order to study changes in skeletal muscle histology and biology.

Functional endpoints in this study include ventilatory gas indices from cardiopulmonary exercise testing, lower body strength testing, grip strength, sit-to-stand, six-minute-walk distance, gait speed, inspiratory muscle strength, and quality of life and physical activity-oriented questionnaires, including the Kansas City Cardiomyopathy Questionnaire, Duke Activity Status Index, and CHAMPS Physical Activity Questionnaire for Older Adults. Body composition is measured with Dual Energy X-ray (DXA) scanning. Skeletal muscle biopsies are completed in the vastus lateralis of the non-dominant leg to assess histology and biologic endpoints.

DETAILED DESCRIPTION:
Despite decades of research, HF remains a common disease that continues to rise in prevalence, particularly among the expanding population of older adults. By virtue of age, older adults are prone to higher incidence of HF and worse clinical consequences. Exercise intolerance and dyspnea are common symptoms that portend poor prognosis, and which erode functional independence and quality of life. Mortality and morbidity also increase significantly as functional capacity declines.

Growing evidence suggests that pathophysiology of central cardiac dysfunction is linked to skeletal muscle pathophysiology. While HF therapeutic guidelines primarily emphasize steps that improve cardiac parameters, and/or volume status, goals to modify HF skeletal muscle myopathy may constitute a vital complementary treatment target.

Ongoing analyses from our pilot VA Merit investigation provide pertinent insights and substantiation. The investigators demonstrated reduced functional capacity (both aerobic and strength) in 31 HF patients (mean age 66 years) compared to 39 age-matched healthy controls (mean age 67). The investigators also showed increased expression of genes signaling ubiquitin-mediated proteolysis in skeletal muscle in relation to decreasing aerobic and strength performance. Consistently, reduced lean muscle mass, as measured by DXA, correlated to the reduced strength indices.

This proposal constitutes a logical progression of this pilot analysis and follows the analytic path the investigators anticipated. Whereas the initial work characterized key skeletal muscle gene expression patterns in association to disease, exercise capacity, and body composition, this study compares the effects of three exercise training regimens (i.e., aerobic vs. combined aerobic and strength vs. inspiratory muscle training [IMT]) each with a unique physiological rationale. The investigators will explore differences in how each training regimen modifies clinical attributes (function/symptoms) as well as skeletal muscle biology that likely underlie these differences. These insights will help identify therapeutic strategies that better suppress injurious disease mechanisms and thereby facilitate improved clinical outcomes and quality of life.

Specific Aims:

a. To assess differences in functional outcomes (peak oxygen utilization [VO2]) and one-repetition max [1RM]) relative to different training regimens: a. Aerobic vs. Aerobic-Strength vs. inspiratory Muscle Training (IMT).

i. Analyses will include assessments of training differences in respect to broader functional parameters (aerobic, strength, inspiration), symptoms, and quality of life.

b. To assess gene expression in relation to the different training regimens.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Heart failure
* Echo in two years
* NYHA class II or III
* Optimal therapy according to AHA/ACC and HFSA HF guidelines; unless documented by a provider for variation.

Exclusion Criteria:

* Major cardiovascular event or procedure within the prior 6 weeks.
* Dementia
* Severe COPD (FEV1<50%),
* End-stage malignancy
* Severe valvular heart disease that would make exercise un safe
* Orthopedic limitation preventing exercise
* Any bleeding disorder that would contraindicate safe exercise
* Women who are pregnant, breastfeeding, or likely to become pregnant within the next 6 months
* Psychiatric hospitalization within the last 3 months
* ICD device with heart rate limits that prohibit exercise assessments or exercise training.

  * Referring physicians will be provided with an opportunity to reprogram devices so that patients can participate.
* Chronic use of oral corticosteroids or medications that affect muscle function.

  * Notably, patients using statins will be eligible, and this will be factored into the randomization and analysis.
* Chronic ETOH or drug dependency shown within the last year

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E. Forman, MD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (2):
- United States (2):
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 65 participants consented to enroll in the study. 45 participants completed a baseline assessment and were randomized to one of the three intervention arms.
  The remaining 20 participants withdrew prior to completing baseline and before being randomized to one of the three intervention arms, so they are not included in this table. Serious adverse events reported after consent but prior to withdrawal for the non-randomized participants are included in a separate group in the adverse events table.
Groups:
- Aerobic Exercise Intervention: Participants completed a 12-week exercise training regimen consisting of aerobic exercise for a minimum of 60 minutes in length three times a week.
- Combined Aerobic and Strength Exercise Intervention: Participants completed a 12-week exercise training regimen consisting of combined aerobic and strength exercise for a minimum of 60 minutes in length three times a week.
- Inspiratory Muscle Training Exercise Intervention: Participants completed a 12-week exercise training regimen consisting of inspiratory muscle training exercise for a minimum of 60 minutes in length three times a week.
Period: Overall Study
Arm/Group | Aerobic Exercise Intervention | Combined Aerobic and Strength Exercise Intervention | Inspiratory Muscle Training Exercise Intervention
Started | 16 | 17 | 12
Completed | 10 | 13 | 11
Not Completed | 6 | 4 | 1
Not completed — Lost to Follow-up | 1 | 2 | 0
Not completed — Withdrawal by Subject | 5 | 2 | 1

BASELINE CHARACTERISTICS:
Population: 65 participants consented to enroll in the study. Baseline demographics were captured for 48 of the participants who consented.
  20 participants who consented to participate withdrew consent prior to completing baseline and prior to randomization. Baseline data were captured for 7 of these 20 participants prior to withdrawal.
  45 participants completed baseline and were randomized to one of the three study arms. Baseline demographics were missing for 4 of these 45 randomized participants.
Groups:
- Consented But Withdrew Pre-randomization: This group includes participants who consented to enroll in the study, but only completed partial or no baseline functional or questionnaire assessments, and then withdrew from the study prior to being randomized. Therefore these participants were not randomly assigned to one of the three study arms, but baseline demographic data were collected after consent and prior to randomization. The baseline demographic data are included here for completion.
- Total: Total of all reporting groups
Arm/Group | Aerobic Exercise Intervention | Combined Aerobic and Strength Exercise Intervention | Inspiratory Muscle Training Exercise Intervention | Consented But Withdrew Pre-randomization | Total
Number analyzed (Participants) | 16 | 13 | 12 | 7 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (7.5) | 67.6 (7.9) | 69.2 (5.0) | 70.7 (9.8) | 69.7 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 16 | 13 | 12 | 7 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 3 | 1 | 0 | 9
  White | 7 | 10 | 10 | 1 | 28
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 1 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Oxygen Uptake (VO2) Peak
Description: a cardiopulmonary exercise test will be performed to determined peak VO2 in ML/KG/Min
Time Frame: baseline and through study completion an average of 14 weeks
Population: Pre and post peak VO2 data available for 33 of 45 randomized participants. Remaining randomized participants did not complete a post assessment so are excluded from the table.
Measure: Mean (Standard Deviation); unit: ML/KG/Min
Arm/Group | Aerobic Exercise Intervention | Combined Aerobic and Strength Exercise Intervention | Inspiratory Muscle Training Exercise Intervention
Number analyzed (Participants) | 10 | 12 | 11
ML/KG/Min
  Baseline | 1778.1 (679.1) | 1228.2 (519.4) | 1393.7 (305.3)
  Follow-up | 1763.6 (736.6) | 1295.4 (499.4) | 1405.9 (370.7)

2. Primary Outcome: One Repetition Maximum- Leg Press
Description: Leg press will be performed on the Keiser Leg press and measured in kilograms (kg)
Time Frame: baseline and through study completion an average of 14 weeks
Population: Data available for 30 of 45 randomized participants who completed both a pre and post assessment.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Aerobic Exercise Intervention | Combined Aerobic and Strength Exercise Intervention | Inspiratory Muscle Training Exercise Intervention
Number analyzed (Participants) | 10 | 11 | 9
kg
  1 Rep Max Leg press baseline | 430.3 (208.6) | 348.2 (143.0) | 421.1 (100.1)
  1 Rep Max Leg press follow-up | 433 (232.7) | 355.5 (160.3) | 409.5 (136.4)

3. Secondary Outcome: Metabolomics
Description: Nitric Oxide Bioavailability (uM) Metabolomics
  The scientific direction of our analyses for this measure has shifted over time. The investigators will pursue RNA seq and metabolomics to provide an unbiased path forward on viable targets in the muscle.
Time Frame: baseline and through study completion an average of 14 weeks
Population: Nitric oxide bioavailability metabolomics data were collected for 23 of the participants at both the baseline and follow-up assessments.
Measure: Mean (Standard Deviation); unit: micrometer (uM)
Arm/Group | Aerobic Exercise Intervention | Combined Aerobic and Strength Exercise Intervention | Inspiratory Muscle Training Exercise Intervention
Number analyzed (Participants) | 5 | 9 | 9
micrometer (uM)
  Baseline Nitric Oxide (uM) | 6.2 (3.7) | 7.7 (2.5) | 7.2 (3.5)
  Follow-up Nitric Oxide (uM) | 5.6 (2.4) | 10.8 (8.9) | 6.6 (3.1)

4. Secondary Outcome: Skeletal Muscle Gene Expression
Description: Skeletal muscle gene expression will be measured in RNA isolated from skeletal muscle biopsy samples via Illumina platform.
  The measure "Number" indicates the number of differentially expressed genes, and units are fold change over baseline. To investigate how the lifestyle interventions impacted gene expression at the mRNA level in skeletal muscles of our research participants we performed high-throughput RNA-Sequencing (Illumina HiSeq paired-end 150 base pairs). Differential gene expression analysis was performed on the RNA-seq. data using DeSEQ2 to determine differentially expressed genes (DEGs) between groups. All DEG analyses were performed using the Wald test (p < 0.05) corrected for multiple comparisons using the Benjamini and Hochberg method.
Time Frame: baseline and through study completion an average of 14 weeks
Population: Skeletal muscle samples were collected for 19 participants who completed both a baseline and follow-up assessment.
Measure: Number; unit: Fold change over baseline
Arm/Group | Aerobic Exercise Intervention | Combined Aerobic and Strength Exercise Intervention | Inspiratory Muscle Training Exercise Intervention
Number analyzed (Participants) | 4 | 7 | 8
Fold change over baseline | 0 | 1 | 1

5. Secondary Outcome: Quality of Life and Daily Function Questionnaires
Description: Participants completed the Kansas City Cardiomyopathy questionnaire (KCCQ) and Duke Activity Status (DASI) Index standardized questionnaires.
  The KCCQ is scored on a scale of 0 to 100 with a higher score representing better health status.
  DASI is a 12-item questionnaire that is scored on a scale of 0 to 58.2, with a higher score representing a higher functional status.
Time Frame: baseline and through study completion an average of 12 weeks
Population: Questionnaire data available for 32 participants who completed both the baseline and 12-week follow-up assessments.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Aerobic Exercise Intervention | Combined Aerobic and Strength Exercise Intervention | Inspiratory Muscle Training Exercise Intervention
Number analyzed (Participants) | 10 | 12 | 10
scores on a scale
  KCCQ Baseline Score | 36 (10.6) | 37.7 (12.0) | 39.5 (16.2)
  KCCQ Follow-up Score | 40 (14.0) | 38 (13.2) | 43 (19.1)
  DASI Baseline Overall Score | 37.3 (14.6) | 34.7 (15.4) | 33.4 (12.2)
  DASI Follow-up Overall Score | 37.3 (15.2) | 32.9 (13.0) | 33.4 (15.9)

6. Secondary Outcome: Community Healthy Activities Model Program for Seniors (CHAMPS) Physical Activity Questionnaire for Older Adults - Frequency Component
Description: Participants completed the Community Healthy Activities Model Program for Seniors (CHAMPS) Physical Activity Questionnaire for Older Adults as part of the Quality of Life and Daily Function study outcome.
  The CHAMPS questionnaire assesses duration and frequency of self-reported weekly physical activities of varying intensities in older adults.
  One component of the CHAMPS score is the frequency per week (i.e. number or count of events per week) that the participant reported that they engaged in all exercise related activities, and the frequency per week that the participant engaged in moderate-vigorous activities.
  The mean frequency of activities per week at baseline and follow-up for each study arm are reported here for the participants who completed both a baseline and follow-up assessment. A higher mean indicates a higher number of exercise-related activities were reported per week.
Time Frame: baseline and through study completion an average of 12 weeks
Population: Questionnaire data available for 32 participants who completed both the baseline and 12-week follow-up assessments. The mean at baseline and 12-week follow-up are reported.
Measure: Mean (Standard Deviation); unit: events per week
Arm/Group | Aerobic Exercise Intervention | Combined Aerobic and Strength Exercise Intervention | Inspiratory Muscle Training Exercise Intervention
Number analyzed (Participants) | 10 | 12 | 10
events per week
  Baseline Mean Frequency of all Physical Activity bouts per week (CHAMPS) | 14.7 (9.2) | 13.6 (9.3) | 9.5 (4.2)
  Follow-up Mean Frequency of all Physical Activity bouts per week (CHAMPS) | 23.5 (10.9) | 22.5 (11.8) | 19.5 (9.1)
  Baseline Mean Frequency of Moderate-Vigorous Physical Activity bouts per week (CHAMPS) | 5.5 (5.6) | 6.3 (4.9) | 3.0 (2.9)
  Follow-up Mean Frequency of Moderate-Vigorous Physical Activity bouts per week (CHAMPS) | 12.1 (8.1) | 10.6 (6.7) | 7.7 (4.9)

7. Secondary Outcome: Community Healthy Activities Model Program for Seniors (CHAMPS) Physical Activity Questionnaire for Older Adults - Duration Component
Description: Participants completed the Community Healthy Activities Model Program for Seniors (CHAMPS) Physical Activity Questionnaire for Older Adults as part of the Quality of Life and Daily Function study outcome.
  The CHAMPS questionnaire assesses duration and frequency of self-reported weekly physical activities of varying intensities in older adults.
  One component of the CHAMPS score is the self-reported duration in hours per week of all exercise-related activities, and duration in hours per week of moderate-vigorous exercise-related activities.
  The mean duration of all exercise-related activities and moderate-vigorous activities in hours per week are reported here for participants in each study arm who completed both the baseline and 12 week follow-up assessments. A higher mean indicates that a longer duration of exercise-related activities in hours per week were reported.
Time Frame: baseline and through study completion an average of 12 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours per week
Arm/Group | Aerobic Exercise Intervention | Combined Aerobic and Strength Exercise Intervention | Inspiratory Muscle Training Exercise Intervention
Number analyzed (Participants) | 10 | 12 | 10
hours per week
  Baseline Mean Duration of all Physical Activity bouts (CHAMPS) | 15.2 (8.1) | 7.7 (4.5) | 5.7 (3.2)
  Follow-up Mean Duration of all Physical Activity bouts (CHAMPS) | 21.8 (15.9) | 14.3 (8.6) | 14.4 (9.6)
  Baseline Mean Duration of Moderate-Vigorous Physical Activity bouts (CHAMPS) | 6.8 (8.5) | 3.5 (2.7) | 1.8 (1.9)
  Follow-up Mean Duration of Moderate-Vigorous Physical Activity bouts (CHAMPS) | 11.6 (11.7) | 7.4 (6.2) | 5.5 (5.4)

8. Other Pre Specified Outcome: Inflammation - C-reactive Protein
Description: Inflammation - C-reactive protein (CRP) will be measured through blood
Time Frame: baseline and through study completion an average of 14 weeks
Population: Data for the C-reactive protein outcome was collected for 28 participants.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Aerobic Exercise Intervention | Combined Aerobic and Strength Exercise Intervention | Inspiratory Muscle Training Exercise Intervention
Number analyzed (Participants) | 8 | 9 | 11
mg/L
  Baseline CRP (mg/L) | 3.3 (1.5) | 3.8 (2.5) | 1.8 (1.6)
  Follow-up CRP (mg/L) | 4.1 (4.1) | 4.2 (3.4) | 2.1 (2.1)

9. Other Pre Specified Outcome: Dual-energy X-ray Absorptiometry
Description: dual-energy x-ray absorptiometry will look at muscle mass change in kg
Time Frame: Baseline and through study completion an average of 14 weeks
Population: 23 randomized participants completed baseline dual-energy x-ray absorptiometry, and 15 of those completed the follow-up scan.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Aerobic Exercise Intervention | Combined Aerobic and Strength Exercise Intervention | Inspiratory Muscle Training Exercise Intervention
Number analyzed (Participants) | 4 | 11 | 8
kg
  Appendicular Lean Mass Baseline | 3.96 (1.14) | 3.08 (0.45) | 3.08 (0.49)
  Appendicular Lean Mass Follow-up: number analyzed (Participants) | 2 | 6 | 7
  Appendicular Lean Mass Follow-up | 8.73 (1.29) | 7.74 (1.28) | 7.72 (0.99)

ADVERSE EVENTS:
Time Frame: After consent through study completion, up to 12 weeks
Description: Serious Adverse Events (SAEs) were reported for participants who consented to the study and were therefore considered enrolled. Some participants experienced an adverse event after consent but prior to completing the full baseline assessments, and withdrew from the study before they were randomized to one of the three intervention arms. For completion, the SAEs reported for these participants are listed in a separate "consented but withdrew pre-randomization" column.
Groups:
- Consented But Withdrew Pre-randomization: Participants who consented to enroll in the study, but only completed partial or no baseline assessments and then withdrew from the study prior to being randomized. These participants were not assigned to one of the three study arms, but had adverse event data that was reported after their consent and prior to withdrawal.
Arm/Group | Aerobic Exercise Intervention | Combined Aerobic and Strength Exercise Intervention | Inspiratory Muscle Training Exercise Intervention | Consented But Withdrew Pre-randomization
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17 | 0/12 | 0/5
Serious Adverse Events (participants affected / at risk) | 10/16 | 3/17 | 5/12 | 5/5
Other Adverse Events (participants affected / at risk) | 0/16 | 0/17 | 1/12 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aerobic Exercise Intervention (N=16) | Combined Aerobic and Strength Exercise Intervention (N=17) | Inspiratory Muscle Training Exercise Intervention (N=12) | Consented But Withdrew Pre-randomization (N=5)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Hospitalization, unrelated to study
Gout (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — ED, unrelated to study
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — ED, unrelated to study
Eye Surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Pre-planned, unrelated to study
Shoulder fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — ED, unrelated to study
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Hospitalization, unrelated to study
Mechanical Fall with Fractures (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Hospitalization, unrelated to study
Acute Heart Failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Hospitalization, unrelated to study
Feeling faint (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Hospitalization, unrelated to study
Acute Heart Failure (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — Hospitalization, unrelated to study
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Referral, unrelated to study
LV thrombus (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Follow-up, unrelated to study
Stomach, Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — ED, unrelated to study
Shoulder pain after fall on ice (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — ED, unrelated to study
Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Hospitalization, unrelated to study
dizziness, SOB, fogginess after medication change (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — ED, unrelated to study
Unknown Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Hospitalization, unrelated to study
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Hospitalization, unrelated to study
Mechanical fall on head (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Hospitalization, unrelated to study
Hypoglycemia (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — ED, unrelated to study
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — ED, unrelated to study
Thigh skin flap removal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Pre-planned, unrelated to study
Lightheadedness after starting new medication (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — ED, unrelated to study
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Hospitalization, unrelated to study
Edema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — ED, unrelated to study
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aerobic Exercise Intervention (N=16) | Combined Aerobic and Strength Exercise Intervention (N=17) | Inspiratory Muscle Training Exercise Intervention (N=12) | Consented But Withdrew Pre-randomization (N=5)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — ED, unrelated to study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/62/NCT03648762/Prot_SAP_000.pdf